CLINICAL TRIAL: NCT06695338
Title: Submerged Vs Non-Submerged Guided Bone Regeneration Simultaneous to Implant Placement.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Germán E. Pardo Perl, DDS, MSc, PhD (Cand), Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER-ECL-2021-10
Record Dates: First submitted 2024-09-29; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Guided Bone Regeneration; Dental Implant; Submerged Regeneration; Bone Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Submerged Approach) (Active Comparator): Standard/Conventional approach in which guided bone regeneration simultaneous to implant placement is leaved submerged under gingival tissue by suturing looking for first intention healing.
  Interventions: Procedure: Guided Bone Regeneration (Submerged)
- Test Group (Non-Submerged Approach) (Experimental): To test approach in which guided bone regeneration simultaneous to implant placement is leaved in a non-submerged manner with second intention healing around an abutment and interproximal suturing.
  Interventions: Procedure: Guided Bone Regeneration (Non-submerged)

INTERVENTIONS:
Procedure: Guided Bone Regeneration (Submerged) — Guided Bone Regeneration by means of bone xenograft and collagen membrane (submerged approach)
  Arms: Control Group (Submerged Approach)
Procedure: Guided Bone Regeneration (Non-submerged) — Guided Bone Regeneration by means of bone xenograft and collagen membrane (Non submerged Approach)
  Arms: Test Group (Non-Submerged Approach)

SUMMARY:
Dental implants are worldwide recognized one of the best manners to replace lost or hopeless prognosis teeth. There are different variables that creates proper conditions for long-term prognosis of implant treatments.

Implant position and surrounding bone around them, have been described in scientific literature to be key factors in the longevity of those treatments.

It has to be defined the "critical bone thickness" around implants. It basically means that implants has to be completely surrounded by bone, that will serve as protection. If the implants are not surrounded by bone, procedures as guided bone regeneration may be performed.

Those procedures can be executed before or simultaneously during the implant placement. In the standard procedure, the simultaneous guided bone regeneration during implant placement requires to leave the implant and the regeneration healing below the gingiva, needing a second surgery for accesing to those implants.

In this randomized controlled trial the hypothesis is to discover if not submerging this regenerations may show the same results than submerged ones.

For that, the objective is to study the different variables around these regeneration to evaluate the performance of non-submerged protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women over 18 years old.

  * Patients requiring single-unit implant restoration in any tooth site of the maxilla and mandible in between teeth.
  * Anticipation of a peri-implant buccal osseous dehiscence by means of a CT imaging (cone-beam computed tomography, CBCT) with a maximum vertical dimension height (VDH) of 50%.
  * Presence of adjacent teeth.
  * Presence of antagonist teeth.
  * Minimum primary stability of 25Ncm.
  * Non-smokers or light smokers (< 10 cigarettes per day).
  * Absence of systemic diseases that could influence the outcome of the therapy (i.e., uncontrolled diabetes mellitus, osteoporosis, biphosphonate medication).
  * Tooth extraction performed at least 4 months before implant placement.
  * Good level of oral hygiene (Plaque Index < 25%) (Löe, 1967)
  * Written informed consent signed.
  * Keratinized mucosa of at least 2mm on the buccal and lingual of the implant.

Exclusion Criteria:

* Implant surgery requiring sinus lift procedure.

  * Previous bone augmentation at the implant site.
  * Active periodontal disease.
  * Acute infection at the rehabilitation site.
  * Long-term non-steroidal anti-inflammatory drug therapy (3 months).
  * Lactating females or currently pregnancy.
  * Severe cognitive or psychiatric disorders.
  * Unwillingness to return for follow-up examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Vertical bone dimensional changes | 0-12months
  Comparison between CBCT images. Vertical bone changes in mm from initial CBCT to 12 months CBCT will be asessed.

SECONDARY OUTCOMES:
Horizontal bone dimensional changes | 0-12 months
  Comparison between CBCT images
Buccal Bone thickness (Dehiscence resolution) | 0-12 months
  Comparison between CBCT images
Marginal Bone Loss (MBL) | 0-12 months
  Comparison between 2d xrays
Peri-implant clinical parameters | 0-12 months
  Clinical variables
Volumetric parameters | 0-12 months
  Comparison between STL's models
PROMs | 0-12 months
  Patient Related Outcomes. (Overall satisfaction from 1-10, Pain perceived from 1-10, Willingness to repeat in case of need from 1-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Uic Barcelona, Barcelona, Spain